CLINICAL TRIAL: NCT01292759
Title: An Evaluation of a New, Non-invasive Monitoring Device in Major Abdominal Surgery Patients
Brief Title: Non-invasive Assessment of Arterial Blood Pressure and Functional Hemodynamic Parameters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Larissa Philippi, Klinik für Anästhesie
Other Study IDs: 837.194.10 (7203)
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2010-07

CONDITIONS: Surgical Procedure, Unspecified
Keywords: stroke volume; cardiac output; validation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cardiac output can be monitored using different invasive devices. Nexfin HD is a new, noninvasive device that uses model flow technology to measure stroke volume and thus computes cardiac output (CO). To evaluate this new device the investigators compared esophageal doppler CO to Nexfin HD CO in patients scheduled for elective abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 80 years old
* Written informed consent obtained

Exclusion Criteria:

* Renal failure
* Heart failure (EF < 25%)
* Peripheral artery occlusion disease
* M. Raynaud
* Rhythms other than sinus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2010-07

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Anaesthesiology der Universitätsmedizin Mainz, Mainz, Germany